CLINICAL TRIAL: NCT06767215
Title: Spasmodic Dysphonia Patients' Perception of Pain With Botulinum Toxin Injections
Brief Title: Dysphonia Pain Perception Following Botulinum Toxin Injections
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Amanda Hu, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: H24-03992
Record Dates: First submitted 2025-01-06; First posted 2025-01-09 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Spasmodic Dysphonia
Keywords: spamodic dysphonia; pain perception; ice compress
MeSH Terms: conditions — Dysphonia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botulinium injection with ice compress (Experimental)
  Interventions: Other: Ice Compress
- Botulium injection without ice compress (Active Comparator)
  Interventions: Other: No ice compress

INTERVENTIONS:
Other: Ice Compress — Ice compress will be applied 5 minutes before butulinium injection
  Arms: Botulinium injection with ice compress
Other: No ice compress — No ice compress will be applied .
  Arms: Botulium injection without ice compress

SUMMARY:
Spasmodic dysphonia (SD) is a chronic voice disorder which can cause a significant decrease in voice related quality of life with no cure. The most common treatment is botox injections in the larynx, with the effect lasting for about 3 months. The procedure is performed in awake, unsedated conditions therefore patients experience pain which in turn affects the tolerance of the procedure. The investigators seek to study whether applying ice compress immediately before the injection would decrease SD patients' perception of pain with botulinum toxin injection. This will be achieved by giving the patients pain questionnaires to complete 10 minutes after the procedure.

DETAILED DESCRIPTION:
Purpose: To determine if ice compress would decrease spasmodic dysphonia patients' perception of pain with botulinum toxin injection.

Hypothesis: Patients will perceive lower levels of pain with applying ice compress.

Justification: There is a lack of data in the available literature on patients' pain perception with botulinum toxin injections and interventions used to decrease pain perception. Applying ice compress (cryotherapy) has strong short-term analgesic effects for various painful conditions, especially in the musculoskeletal system, like acute sports injury, post-op orthopaedic surgery, and dental conditions. However, cryotherapy has not been used much in otolaryngology. This study will provide insights on possible use of cryotherapy in this field.

Objectives: The investigators aim to evaluate if there is any significant difference in pain perception of patients who undergo botulinum injection with application of ice compress prior to the injection.

Research Design: This will be a prospective unblinded randomized controlled study with cross over design. Adductor SD patients will be recruited from the UBC Pacific Voice Clinic run by PI, Dr. Amanda Hu. Interested patients will be provided more information regarding the study and will be consented during their clinic visit. Recruited patients will receive transcutaneous transcricothyroid injection of botulinum toxin with alternating use of no anesthesia (control) or ice compress (intervention) in two consecutive laryngeal injections, which most patients receive every 3-4 months. Intervention for the purpose of this study will be applying ice compress to neck for 5 minutes prior to botulinum toxin injection. Ten minutes after the procedure, patients will complete the short form McGill Pain Questionnaire. Pain scores will be compared for each participant with ice compress and without the ice compress. the investigators will also collect other factors that may affect pain from the medical charts as follows: Age, gender, body mass index, employment status (employed vs unemployed), Voice Handicap Index, opioid usage (yes/no), psychiatric medications (yes/no), chronic pain history (yes/no), duration of diagnosis, botox injection dose, bilateral/unilateral, first injection vs subsequent injection, professional voice user (yes/no), ever smoker (current and former vs never), completion of procedure (yes/no). The investigators will asses if there is a significant relationship between any of these factors and SD patients' pain perception.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (18 years old and older) with adductor spasmodic dysphonia who present to the UBC Pacific Voice clinic for botulinum toxin injections.

Exclusion Criteria:

1. Patients with abductor or mixed spasmodic dysphonia
2. Patients who do not speak English
3. Patients without the mental capacity to complete the study
4. Patients less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Pain score | 10 min after the injection.
  Patients will be asked to complete Short Form McGill Questionnaire (SF-MPQ) pain questionnaire that has a visual acuity pain (VAS) score integrated in it to obtain pain level. The minimum and maximum levels of scale are 0 and 100 and higher scores mean worse pain levels.

IPD SHARING:
Plan to Share IPD: Undecided